CLINICAL TRIAL: NCT07050654
Title: Studio Della Motivazione All'Esercizio Fisico in modalità Social Dual-task in Ambiente di realtà Virtuale Non Immersiva" Nell'Ambito Del Progetto ActivE3 - Everyone, Everywhere, Everyday "Rif. 2021-0612 - CUP C13C21000200005
Brief Title: Motivation While Doing Physical Exercise in a Social Dual-task Virtual Environment
Acronym: ActivE3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto di Sistemi e Tecnologie Industriali Intelligenti per il Manifatturiero Avanzato (Other)
Collaborators: IRCCS Eugenio Medea (Other); Centro Riabilitativo Villa Beretta (Unknown); Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: L2-245
Record Dates: First submitted 2025-06-03; First posted 2025-07-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteer; Stroke; COPD; Cerebral Palsy
MeSH Terms: conditions — Stroke; Pulmonary Disease, Chronic Obstructive; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-player mode: Social Bike (Experimental): The participants engage in cognitive exercises while cycling through two virtual scenarios: a park and an urban environment. Three cognitive tasks are available to perform while cycling. Each task has been designed to focus on one or more cognitive abilities and try to reproduce activities and situations of daily living as much as possible.
  Each exercise is performed in couple, collaborating or competing with another peer. Participants communicate with each other thanks to a voice chat.
  In the case of competitive gameplay, both participants are expected to perform the same task and respond to the same stimuli. Each participant can view their own score as well as the score of their opponent.
  In the case of collaborative gameplay, the system allows participants to view the same environment and engage in the same task. However, participants take turns playing for a fixed number of seconds, determined by the therapist.
  Interventions: Device: Dual-task cycling
- Single-player mode (Active Comparator): The same dual-task exercises described for the social modality can be played also in a single-player mode. Participants perform the cognitive task autonomosly and increase only their personal score.
  Interventions: Device: Dual-task cycling

INTERVENTIONS:
Device: Dual-task cycling — Pairs of participants are formed, who will be the SocialBike players; these pairs consist of users from the same center. The two players are in the same room where two replicas of the SocialBike system are installed.
  The participants can each view, on their own screen, the virtual scenario, either a park or a city environment. Movement within these VR environments is synchronized with the patient's actual pedaling speed, measured in revolutions per minute (RPM) from the cycle ergometer. Movement occurs along a predefined path. The participant's heart rate will always be monitored.
  The therapist chooses the optimal ergometer workload, the type of exercise, and social/single-player mode. Each session (either single- or multi-player mode) lasts 10 minutes. The available exercise are: "Find the intruder" (go/no-go task); "Prepare your Meal" (spatial attention); "Watch the road" (working memory).

SUMMARY:
The goal of this interventional study is to assess the difference in participants' motivation while performing a virtual reality-based dual-task exercise in a single-player vs. multi-player modality. The populations involved are the following: healthy young adults (14-18 ys.); children and adolescents (12-17 ys.) with motor disorders; older adults with neurological or respiratory conditions. The main questions it aims to answer are:

Is a "social" virtual environment better in promoting motivation to perform physical exercise? Is a "social" virtual environment better in promoting involvement, perceived social inclusion, and exercise performance?

Forty participants will test the single-player and the multi-player scenarios in a single-session and will rate their experiences with subjective questionnaires. A subgroup of participants (12) will use the multi-player system for 3 weeks/3 times a week.

ELIGIBILITY:
Inclusion Criteria:

* For IRCCS E. Medea: patients 12 years and older with neuromotor pathologies;
* For Villa Beretta: adults with neurological pathologies;
* For INRCA Casatenovo: patients with chronic respiratory diseases, clinical stability for at least 4 weeks;
* Healthy volunteers: healthy students aged 14-18 years.

Exclusion Criteria:

* Absence of appropriate cognitive abilities to interact with virtual reality software;
* Presence of severe sensory deficits (visual acuity, auditory perception) such as to interfere with the administration of the proposed activities;
* Poor trunk control or physical limitations (excessive spasticity or joint limitations) that impair the safe performance of the pedaling activity. Presence of epilepsy or treatment with antiepileptic drugs, where the physician highlights contraindications;
* Participation in other standardized rehabilitation protocols involving lower limbs and walking.

Specifically, for INRCA Casatenovo:

* clinical instability (pH <7.35, hemodynamic instability, resting tachypnea);
* acute exacerbations in the month prior to enrollment;
* cognitive impairment such that participation in rehabilitation activities is impaired (Mini Mental State Examination < 24);
* cardiovascular decompensation NYHA (New York Heart Association) class III and IV;
* major cardiac arrhythmias;
* active solid or hematologic neoplasms;
* recent myocardial infarction (< 6 months);
* orthopedic clinical conditions that interfere with exercise.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Motivation | Day 1 - at the end of the test with Condition 1 (single- or multi-player); Day 1 - at the end of the test with Condition 2 (multi- or single-player). At the end of the 4th and the 8th sessions for the participants performing 3 weeks of training.
  Situational Motivation Scale (SIMS; Guay et al. 2000). This questionnaire is composed of 16 items to be rated with a Likert scale going from 1 (corresponds not all) to 7 (corresponds exactly). Items are grouped in four different subscale (Intrinsic Motivation, Identified Regulation, External Regulation, Amotivation). Each subscale score can vary between 1 (minimum) and 7 (maximum).

SECONDARY OUTCOMES:
Usability | Day 1
  System Usability Scale (Brooke, 1996) - The scale ranges from 0 to 100. Higher scores indicate better usability.
  Ratings can be described as follows: "Excellent" (85-100); "Good" (70-84); "Average" (50-69); "Poor" (<50).
Involvement | Day 1 - at the end of the test with Condition 1 (single- or multi-player); Day 1 - at the end of the test with Condition 2 (multi- or single-player). At the end of the 4th and the 8th sessions for the participants performing 3 weeks of training.
  Game Experience Questionnaire (GEQ) (IJsselsteijn, et al., 2013)- GEQ is composed of several subscales: Competence, Sensory and Imaginative Immersion, Flow, Tension/Annoyance, Challenge, Negative Affect, Positive Affect.
  Each subscale ranges from 0, which means "Not at all", and 4, which means "Extremely". Higher score corresponds stronger experience in that dimension.
Perceived social inclusion | Day 1 - at the end of the test with Condition 1 (single- or multi-player); Day 1 - at the end of the test with Condition 2 (multi- or single-player). At the end of the 4th and the 8th sessions for the participants performing 3 weeks of training.
  ad-hoc question; the question will address how much participants feel included while performing the physical activity. The answer ranges from 0 "not at all" to 4 "completely included".
Game and physical performance | Data are stored automatically by the system each time the application is launched. Outcomes data are collected during each session of SocialBike use, i.e., during the single-sessions and each session of the 3 weeks of training.
  The system automatically stores a file containing each player game and physical data for the session. In particular, the file will contain the exercise information: scenario, duration, task performed, level of difficulty, game mode (collaborative/competitive). In terms of performance, the following outcomes will be collected: average speed [revolutions per minute], average heart rate [beats per minute], personal score in the cognitive task [# points collected], final score in [# points collected by the two players if collaborative, equal to personal if competitive].
Endurance | At the baseline; at the end of the 8th session (only for participants performing the 3 weeks of training).
  Assisted 6-minute cycling test (A6MCT)
Physical activity inclination | At the baseline; at the end of the 8th session (only for participants performing the 3 weeks of training).
  Ad-hoc question; the question will address how much participants are motivated in performing physical activity. The answer ranges from 0 "not at all" to 4 "extremely motivated".
Attitude toward technology | At the baseline; at the end of the 8th session (only for participants performing the 3 weeks of training).
  Ad-hoc question; the question will address how much participants feel at ease while interacting with technology. The answer ranges from 0 "not at all" to 4 "extremely at ease".

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - IRCCS E. Medea, Bosisio Parini, LC
  - IRCCS INRCA Casatenovo, Casatenovo, LC
  - Villa Beretta Rehabilitation Clinic - Valduce Hospital, Costa Masnaga, LC
  - CNR-STIIMA - Lecco, Lecco, Lecco

IPD SHARING:
Plan to Share IPD: No